CLINICAL TRIAL: NCT03316326
Title: A Phase II Study of S-1, Irinotecan, and Oxaliplatin in Locally-Advanced Pancreatic Cancer (SIROX Study) - Followed by Curative Surgery and Adjuvant Chemotherapy
Brief Title: S-1, Irinotecan, and Oxaliplatin in Locally-Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201610076MIPB
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — titanium silicide; S 1 (combination); Oxaliplatin; Irinotecan

STUDY DESIGN:
Intervention Model Description: Simon's two-stage optimum design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIROX (Experimental): Tegafur-gimeracil-oteracil potassium, irinotecan, oxaliplatin combination
  Interventions: Drug: Tegafur-gimeracil-oteracil potassium; Drug: Oxaliplatin; Drug: Irinotecan

INTERVENTIONS:
Drug: Tegafur-gimeracil-oteracil potassium — 40 mg bid, D1-14
  Other Names: TS-1; S-1
Drug: Oxaliplatin — 85 mg/m2, D1
  Other Names: Oxalip
Drug: Irinotecan — 150 mg/m2, D8
  Other Names: Irino

SUMMARY:
This phase II clinical trial will enroll patients with newly-diagnosed locally-advanced pancreatic adenocarcinoma and adopt the Simon's two-stage optimum design. After 4 cycles of SIROX regimen, patients will proceed to curative resection.

DETAILED DESCRIPTION:
This phase II clinical trial will enroll patients with newly-diagnosed locally-advanced pancreatic adenocarcinoma and adopt the Simon's two-stage optimum design. After 4 cycles of SIROX regimen, patients will proceed to curative resection. The primary endpoint of this study is resection rate after neoadjuvant chemotherapy. The first stage will enroll 18 patients. We will go into the second stage if at least 2 patients in stage I become resectable after treatment. There will be at most 35 patients enrolled. Based on this trial, we anticipate that the SIROX regimen has comparable response rate and resection rate but lower toxicities comparing to FOLFIRINOX.

ELIGIBILITY:
Inclusion Criteria:

1. histologically or cytologically proven pancreatic adenocarcinoma
2. newly diagnosed, unresectable, locally-advanced pancreatic cancer
3. no potential of R0 resection at diagnosis
4. presence of measurable pancreatic lesion, which must meet the criteria of being ≥ 10 mm in at least one dimension by conventional CT/MRI
5. age between 20 and 79 years at registration
6. ECOG performance status (PS) of 0 or 1
7. adequate major organ functions
8. ability to take the oral study medication (S-1)
9. no clinically significant abnormal ECG findings within 28 days (4 weeks) prior to registration
10. voluntarily signed the written informed consent form

Exclusion Criteria:

1. pulmonary fibrosis or interstitial pneumonitis diagnosed within 28 days prior to registration
2. presence of diarrhea ≥ CTCAE v.4.03 grade 2
3. concomitant active infection
4. significant co-morbid medical conditions, including, but not limited to , heart failure, renal failure, hepatic failure, hemorrhagic peptic ulcer, mechanical or paralytic ileus, or poorly controlled diabetes
5. moderate or severe ascites or pleural effusion that requires drainage
6. prior or concurrent malignancies within the last 3 years, with the exception of carcinoma in situ of the cervix, or basal type skin cancer
7. concomitant treatment with flucytosine, phenytoin or warfarin
8. peripheral neuropathy grade of 2 or higher
9. known Gilbert syndrome or homozygosity for UGT1A1 promoter TA repeats prone to high risk of drug toxicity (screening of UGT1A1 genotype will NOT performed routinely before study)
10. pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential. Patients of childbearing age should have effective contraception for both the patient and his or her partners during the study period
11. severe mental disorder
12. judged ineligible by physician for participation in the study due to safety concern

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
resection rate | 3 years
  patients with R0 or R1 resection of the primary tumor after study chemotherapy/patients receiving at least one dose of study chemotherapy

SECONDARY OUTCOMES:
response rate (RR) | 3 years
  RR of SIROX
Overall survival (OS) | 4 years
  OS of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wen Tien, M.D., Ph. D., Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT03316326/Prot_SAP_000.pdf